CLINICAL TRIAL: NCT01896830
Title: Safety and Immunogenicity of a Clostridium Difficile Toxoid Vaccine Administered to Healthy Adult Subjects Aged 40 to 75 Years in Japan
Brief Title: Study of a Candidate Clostridium Difficile Toxoid Vaccine in Healthy Adult Subjects Aged 40 to 75 Years in Japan
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDI19 (DFI13360); U1111-1127-7547 (Other: WHO)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile infection; Clostridium difficile Toxoid Vaccine
MeSH Terms: conditions — Clostridium Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccine Group (Experimental): Participants will receive the candidate C. difficile toxoid vaccine
  Interventions: Biological: Clostridium difficile Toxoid Vaccine
- Placebo Group (Placebo Comparator): Participants will receive a placebo vaccine
  Interventions: Biological: 0.9% normal saline

INTERVENTIONS:
Biological: Clostridium difficile Toxoid Vaccine — 0.5 mL, intramuscular
  Arms: Vaccine Group
Biological: 0.9% normal saline — 0.5 mL, intramuscular
  Other Names: NaCl
  Arms: Placebo Group

SUMMARY:
The aim of the study is to evaluate a candidate C. difficile Toxoid Vaccine in the Japanese population.

Primary objectives:

* To describe the safety profile of all subjects who receive at least 1 injection
* To describe the immunogenicity to toxin A and toxin B in all subjects from serum samples obtained on Days 0, 14, 30, and 60.

DETAILED DESCRIPTION:
Participants will be randomly assigned to receive the vaccine or placebo on the selected schedule. Safety parameters, solicited injection site and systemic reactions will be collected for 6 days after each injection; unsolicited adverse events including serious adverse events will be collected up to Day 60 post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects aged 40 to 75 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination)
* Participation in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination, except for influenza (seasonal or pandemic) and pneumococcal vaccine.
* Planned receipt of any vaccine between study vaccinations and in the 4 weeks following the last trial vaccination, except for influenza (seasonal or pandemic) and pneumococcal vaccines
* Previous vaccination against C. difficile with either the trial vaccine another vaccine, or monoclonal antibodies
* Self-reported current or prior Clostridium difficile infection (CDI) episode
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Known systemic hypersensitivity to any of the vaccine components (including aluminum hydroxide, sodium citrate,sucrose, formaldehyde, sodium chloride), or history of a life-threatening reaction to a vaccine containing any of the same substances
* Known medical history or concomitant disease of thrombocytopenia
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Subjects who have any history of intestinal diverticular bleeding
* Subjects who have had surgery within the past three months for Gastro-Intestinal malignancy
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 37.5°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Subject who has concomitant disease that, according to investigator's/sub-investigator's judgment, would adversely affect the safety of the subject in the study, e.g., cardiovascular disease, renal disease, hepatic disease, hematologic disease, and/or growth impairment
* Subject with a past history of convulsions
* Subject ineligible for participation in the study according to the investigator's/sub-investigator's judgment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Solicited Injection Site Reactions, Solicited Systemic Reactions, Unsolicited Systemic Reactions, and Serious Adverse Events Occurring Throughout the Trial | Day 0 up to Day 60 post-vaccination
  Solicited injection site reactions: Pain, Redness, and Swelling. Solicited systemic reactions: Fever (temperature), Headache, Malaise, Myalgia, and Arthralgia.
Serum antibody concentrations to toxins A and B, measured by enzyme-linked immunosorbent assay (ELISA) | Day 0 pre-vaccination, Days 14, 30 and 60 post-vaccination
  Serum antibody concentrations to toxins A and B will be measured by enzyme-linked immunosorbent assay (ELISA)
Serum antibody titers against toxins A and B, measured by toxin neutralizing assay | Day 0 pre-vaccination, Days 14, 30 and 60 post-vaccination
  Serum antibody titers against toxins A and B will be measured by toxin neutralizing assay (TNA)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur K.K
Locations (1):
- Osaka, Japan

REFERENCES:
- [Result] Matsuoka O, Patel DM, Sasaki S, Oka H, Sasaki T, Pietrobon PJ, Laot T, Bouckenooghe A, Menezes J, de Bruyn G. Safety and immunogenicity of Clostridium difficile toxoid vaccine in Japanese adults. Hum Vaccin Immunother. 2018 Feb 1;14(2):322-328. doi: 10.1080/21645515.2017.1395538. Epub 2017 Dec 6. PMID 29116880